CLINICAL TRIAL: NCT05279586
Title: Secondary Prophylaxis of Overt Hepatic Encephalopathy in Cirrhosis: a Randomized Controlled Trial of Colistin Versus Lactulose
Brief Title: Secondary Prophylaxis of Hepatic Encephalopathy in Cirrhotic Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Madonna Magdy Fahmy (Other)
Responsible Party: Sponsor-Investigator, Madonna Magdy Fahmy, Principal Investigator, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: encephalopathy prophylaxis
Record Dates: First submitted 2022-02-09; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Lactulose; Colistin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients that will receive lactulose (Active Comparator): Cirrhotic patients who were recovered from HE will be randomized into lactulose group receiving 30-60 ml of lactulose orally in 2 or 3 divided doses so that patient passed 2-3 semisoft stools per day
  Interventions: Drug: lactulose
- patients that will receive colistin (Active Comparator): colistin group receiving colistin sulfate 1.5 million I.U. tablet orally twice
  Interventions: Drug: colistin

INTERVENTIONS:
Drug: lactulose — all interventions are used in secondary prophylaxis in cirrhotic patients
  Other Names: duphlac
  Arms: patients that will receive lactulose
Drug: colistin — all interventions are used in secondary prophylaxis in cirrhotic patients
  Arms: patients that will receive colistin

SUMMARY:
The aim of this study is to compare the efficacy and safety of colistin versus lactulose for secondary prophylaxis of overt hepatic encephalopathy in patients with liver cirrhosis.

DETAILED DESCRIPTION:
Hepatic encephalopathy (HE) is a reversible neuropsychiatric changes, it occurs in 30%-45% of cirrhotic patients during their life. Once HE is developed, the 1-year mortality exceeds 60%. The high morbidity and mortality combined with the costs underline the importance of effective treatment and prevention of HE.

The exact pathogenesis of HE is still unknown but ammonia is known to play a key role. Strategies to prevent and treat HE aims at reducing the production and absorption of gut derived neurotoxins, particularly ammonia, mainly through bowel cleansing, non absorbable disaccharides and non -absorbable antibiotics.

Patients with previous episode of overt HE, have a 40% cumulative risk of recurrence at 1 year. Because recurrent episodes of HE are associated with increased health care burden, poor prognosis, and risk of death, prevention of the recurrence of HE should be considered in each patient.

After an episode of overt HE has resolved, patients with cirrhosis should receive secondary prophylactic therapy for an indefinite period of time or until they undergo liver transplantation. Lactulose is considered the first line for secondary prophylaxis of overt HE while rifaximin is add-on therapy to lactulose.

Non-absorbable disaccharides like lactulose acts as both osmotic laxative, and gut acidifying agent reducing the production and the absorption of ammonia from the intestines by changing the gut microbiota. However, side effects of lactulose therapy including excessively sweet taste and gastrointestinal side effects such as abdominal pain, bloating, flatulence, severe and unpredictable diarrhea possibly leading to dehydration result in frequent non-adherence in clinical practice. Lactulose non-adherence, reported as a factor in 39% of hospital admissions, was the single most frequent precipitant of overt HE .

Rifaximin is a non-absorbable antibiotic with low systemic absorption, broad antimicrobial spectrum, and low frequency of side effects. It has a place in prevention of recurrence of HE when lactulose alone fails. However, the accessibility of rifaximin may be limited by its high cost.

Colistin sulfate is a polymyxin antibiotic which is active against aerobic gram-negative bacteria including most enterobacteria except Proteus. It is poorly absorbed from the gastrointestinal tract. Colistin sulfate being not systemically absorbed is used orally for bowel decontamination and treatment of intestinal infections.

Oral colistin is used for peri-operative selective decontamination of digestive tract in elective colorectal cancer patients in combination with tobramycin and amphotericin B. Also, combining oral colistin with ciprofloxacin has been effective in the prevention of Gram-negative sepsis in neutropenic patients without the emergence of significant resistance. However, no study up till now focuses on the use of oral colistin in the secondary prophylaxis of hepatic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* • Age >18 years.

  * Patients with liver cirrhosis and previous history of recovery from hepatic encephalopathy.

Exclusion Criteria:

* • History of taking lactulose in past 7 days

  * Patients on secondary prophylaxis for spontaneous bacterial peritonitis
  * Patients on psychoactive drugs, such as antidepressants or sedatives
  * Previous transjugular intrahepatic portosystemic shunts or shunt surgery
  * Significant comorbid illness such as heart, respiratory, or neurological disease such as Alzheimer's disease and Parkinson's disease
  * Hepatocellular carcinoma or other neoplasias that could shorten life expectancy
  * Recent infection or antibiotic use within last 6 weeks
  * Recent gastrointestinal bleeding in the past 6 weeks
  * Renal insufficiency, myasthenia gravis.
  * Hypersensitivity to colistin sulfate.
  * Pregnancy or lactation
  * Alcohol intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Development of overt hepatic encephalopathy | 6 months
  Number of Participants with Development of overt hepatic encephalopathy encephalopathy according to West Haven criteria

SECONDARY OUTCOMES:
Health related quality of life | 6 months
  HRQOL assessment using chronic liver disease questionnaire (higher score equates to worse quality of life)